CLINICAL TRIAL: NCT00659165
Title: Exploration of the Weight Neutral Effects of Insulin Detemir Compared to Insulin Glargine: A Measure of Satiety and Calories Consumed in Type 1 Diabetes
Brief Title: Insulin Detemir Compared to Insulin Glargine: Appetite and Calories Consumed in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: UNM HRRC # 08-043
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; insulin dependent diabetes; diabetes mellitus; detemir; levemir; glargine; lantus; insulin; appetite; satiety; centrally acting mediators of satiety; three factor eating questionnaire; PYY; ghrelin; leptin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Detemir (Experimental): Insulin Detemir
  Interventions: Drug: Insulin Detemir
- Insulin Glargine (Experimental): Insulin Glargine
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Detemir — Subjects will be given a dose of detemir equivalent to their current long acting insulin regimen. Study insulin will be injected subcutaneously at 8 AM and 8 PM for at least 3 weeks.
  Other Names: Levemir
  Arms: Insulin Detemir
Drug: Insulin Glargine — Subjects will be given a dose of glargine equivalent to their current long acting insulin regimen. Study insulin will be injected subcutaneously at 8 AM and 8 PM for at least 3 weeks.
  Other Names: Lantus
  Arms: Insulin Glargine

SUMMARY:
Patients with diabetes treated with insulin often gain weight, which may deter patients from adhering to insulin treatment. Detemir is one type of long acting insulin approved by the Food and Drug Administration for use in people with diabetes. It is similar to other long acting insulins (Neutral Protein Hagedorn [NPH], glargine) except that it has been associated with less weight gain compared to other types of insulin. The reasons for this are still unclear. One possibility is that detemir insulin acts differently than do other insulins in affecting how diabetic patients eat meals. The purpose of this study is to determine whether appetite and calories eaten during a meal are affected by the type of insulin used to treat diabetes. This is a pilot study which means we are gathering preliminary information to determine if a larger study can be done.

DETAILED DESCRIPTION:
Insulin detemir is a neutral, soluble long acting insulin analog with weight neutral properties. In limited studies, it has been shown to result in less weight gain in type 1 and type 2 diabetics compared with other long acting insulin formations. A possible mechanism for its weight neutrality is the fatty acid chain that may allow for improved central nervous system activity and effects on satiety. The primary objective of this study is to determine if patients with type 1 diabetes consume fewer calories when allowed to eat to satiety while treated with insulin detemir compared to insulin glargine. Secondary objectives are 1) subject responses on validated satiety scales and food diaries, 2) bioelectrical impedance analysis, 3) resting energy expenditure on indirect calorimetry/metabolic cart measurement, and 4) centrally acting mediators of satiety measured in the serum (Peptide YY [PYY], ghrelin, leptin).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Treated with long-acting and meal time insulin therapy for at least 2 years
* Ages 18 to 60 years of age
* Glycosylated hemoglobin value between 7 - 9 mg/dL
* C-peptide value less than 1.0 pmol/ml 90 minutes after oral Boost Plus administration.

Exclusion Criteria:

* Advanced complications of diabetes (nephropathy, retinopathy, significant neuropathy, coronary artery disease)
* Severe medical illness or medical conditions including congestive heart failure, angina, liver failure or renal failure
* Pregnancy
* Alcohol or drug abuse or dependence within three months of study entry
* Less than 50 % agreement on 50-item Food Questionnaire with the Food Array "buffet style" study meal.
* Women of child-bearing age not adhering to the following contraceptive methods: oral contraceptives, barrier methods including condoms or diaphragm, or abstinence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burge, M.D., Principal Investigator — University of New Mexico, Department of Internal Medicine, Division of Endocrinology; Stephen Mitchell, D.O., Study Director — University of New Mexico, Department of Internal Medicine, Division of Endocrinology
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Bush MA. Intensive diabetes therapy and body weight: focus on insulin detemir. Endocrinol Metab Clin North Am. 2007 Aug;36 Suppl 1:33-44. doi: 10.1016/s0889-8529(07)80006-5. PMID 17881330
- [Background] Drugdex System:Klasko RK: Detemir. Drugdex System. Thomson Micromedex, Greenwood Village, Colorado (2007).
- [Background] Hermansen K, Davies M. Does insulin detemir have a role in reducing risk of insulin-associated weight gain? Diabetes Obes Metab. 2007 May;9(3):209-17. doi: 10.1111/j.1463-1326.2006.00665.x. PMID 17391147
- [Background] Wynne K, Stanley S, McGowan B, Bloom S. Appetite control. J Endocrinol. 2005 Feb;184(2):291-318. doi: 10.1677/joe.1.05866. PMID 15684339
- [Background] Tahbaz F, Kreis I, Calvert D. An audit of diabetes control, dietary management and quality of life in adults with type 1 diabetes mellitus, and a comparison with nondiabetic subjects. J Hum Nutr Diet. 2006 Feb;19(1):3-11. doi: 10.1111/j.1365-277X.2006.00668.x. PMID 16448469
- [Background] Cruz AF, Calle-Pascual AL; Diabetes and Nutrition Study Group, Spanish Diabetes Association. Diabetes Nutrition and Complications Trial: Trends in nutritional pattern between 1993 and 2000 and targets of diabetes treatment in a sample of Spanish people with diabetes. Diabetes Care. 2004 Apr;27(4):984-7. doi: 10.2337/diacare.27.4.984. No abstract available. PMID 15047660
- [Background] Toeller M, Buyken AE, Heitkamp G, Cathelineau G, Ferriss B, Michel G; EURODIAB IDDM Complications Study Group. Nutrient intakes as predictors of body weight in European people with type 1 diabetes. Int J Obes Relat Metab Disord. 2001 Dec;25(12):1815-22. doi: 10.1038/sj.ijo.0801816. PMID 11781763
- [Background] Wilding JP. Neuropeptides and appetite control. Diabet Med. 2002 Aug;19(8):619-27. doi: 10.1046/j.1464-5491.2002.00790.x. PMID 12147141
- [Background] McDuffie JR, Riggs PA, Calis KA, Freedman RJ, Oral EA, DePaoli AM, Yanovski JA. Effects of exogenous leptin on satiety and satiation in patients with lipodystrophy and leptin insufficiency. J Clin Endocrinol Metab. 2004 Sep;89(9):4258-63. doi: 10.1210/jc.2003-031868. PMID 15356018
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Pieber TR, Treichel HC, Hompesch B, Philotheou A, Mordhorst L, Gall MA, Robertson LI. Comparison of insulin detemir and insulin glargine in subjects with Type 1 diabetes using intensive insulin therapy. Diabet Med. 2007 Jun;24(6):635-42. doi: 10.1111/j.1464-5491.2007.02113.x. Epub 2007 Mar 22. PMID 17381500
- [Background] de Graaf C, Blom WA, Smeets PA, Stafleu A, Hendriks HF. Biomarkers of satiation and satiety. Am J Clin Nutr. 2004 Jun;79(6):946-61. doi: 10.1093/ajcn/79.6.946. PMID 15159223
- [Background] Wynne K, Bloom SR. The role of oxyntomodulin and peptide tyrosine-tyrosine (PYY) in appetite control. Nat Clin Pract Endocrinol Metab. 2006 Nov;2(11):612-20. doi: 10.1038/ncpendmet0318. PMID 17082808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sporadic Newspaper advertisement, Albuquerque Journal, July 2008-July 2010.
Pre-assignment Details: Three weeks of treatment with each insulin (glargine, detemir) in random order, double blind assignment. Doses of glargine and detemir were equivalent and were based upon existing long acting insulin doses. Doses were titrated up to achieve target fasting glucose < 150 mg/dl. Both long acting insulins were given once daily before breakfast.
Groups:
- Insulin Detemir: These people receive insulin detemir first, then insulin glargine. All subjects received three weeks of therapy with their assigned insulin prior to overnight admission for study.
- Insulin Glargine: These people receive insulin glargine first, then insulin detemir. All subjects received three weeks of therapy with their assigned insulin prior to overnight admission for study.
Period: Overall Study
Arm/Group | Insulin Detemir | Insulin Glargine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir | Insulin Glargine | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants] — Data for all enrolled subjects in this crossover study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 5 | 10
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Data for all enrolled subjects.
  years | 37 (14) | 33 (8) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Calories Consumed After Fast.
Description: Total energy ingested following the 24 hour fast.
Time Frame: Measured after a 24 hour fast, after treatment with study insulin for at least 3 weeks
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Insulin Detemir | Insulin Glargine
Number analyzed (Participants) | 10 | 10
kcal | 1418 (636) | 1357 (576)

ADVERSE EVENTS:
Arm/Group | Insulin Detemir | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No